CLINICAL TRIAL: NCT07374380
Title: Effect of a Nurse-Led Early Mobilization Protocol on Colorectal Surgery Patients: A Randomized Controlled Trial
Brief Title: Nurse-Led Early Mobilization After Colorectal Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Nebihat Tekin, Clinical Nurse, RN, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 25-12T/49
Record Dates: First submitted 2026-01-06; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Surgery; Early Mobilization; Postoperative Care; Postoperative Recovery
Keywords: colorectal surgery; early mobilization; Nurse-Led Intervention

STUDY DESIGN:
Masking Description: Blinding of participants and care providers is not feasible; however, data analysis will be performed by a statistician blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse-Led Early Mobilization Protocol (Experimental): Participants in the intervention group will receive a structured nurse-led early mobilization protocol, developed in accordance with evidence-based guidelines and current literature, in addition to standard postoperative care. As part of the protocol, patients will receive preoperative education regarding the purpose, benefits, and process of early mobilization, along with a postoperative mobilization brochure. In the postoperative period, mobilization will be initiated within the first 6-8 hours in clinically stable patients under nurse supervision. Mobilization activities will progress gradually, including in-bed exercises, sitting, assisted standing, and walking, with daily walking targets increased on postoperative days 0.-3. All mobilization activities will be delivered by nurses and documented using a standardized mobilization monitoring chart.
  Interventions: Other: Nurse-Led Early Mobilization
- Standard Mobilization Care (Active Comparator): Participants in the control group will receive standard postoperative mobilization care routinely provided in the institution. Mobilization activities will be performed according to existing clinical practices, and no structured or protocol-based nurse-led early mobilization program will be implemented. Participants in the control group will continue to receive usual nursing care without any disadvantage or additional risk in terms of patient care.
  Interventions: Other: Standard Mobilization Care

INTERVENTIONS:
Other: Nurse-Led Early Mobilization — 1. Preoperative Period Patients will receive verbal education regarding the purpose, benefits, and process of early mobilization.
     To support this education, a Postoperative Mobilization Information Brochure prepared by the researchers will be provided to the patient and their caregiver.
  2. Postoperative Day 0 Within the first 6-8 hours after surgery, vital signs will be monitored, and mobilization will be initiated in clinically stable patients under nurse supervision.
  2.1. In-Bed Activities (Postoperative Hour 5)
  The following lower-extremity exercises will be performed:
  Ankle dorsiflexion and plantar flexion Toe movements Leg extension without knee flexion Circular foot movements Each exercise will be performed 5-10 repetitions. The patient will then be positioned in an upright sitting position in bed. 2.2. First Standing and Ambulation (Postoperative Hours 6-8) Vital signs will be assessed. The patient will be assisted to sit at the bedside for 1-2 minutes under nurse
  Arms: Nurse-Led Early Mobilization Protocol
Other: Standard Mobilization Care — Participants in the control group will receive standard postoperative mobilization care routinely provided in the institution. Mobilization activities will be performed according to existing clinical practices, and no structured or protocol-based nurse-led early mobilization program will be implemented. Participants in the control group will continue to receive usual nursing care without any disadvantage or additional risk in terms of patient care.
  Arms: Standard Mobilization Care

SUMMARY:
This study was designed to evaluate the effectiveness of a nurse-led early mobilization protocol on postoperative recovery outcomes in patients undergoing elective colorectal surgery. The outcomes assessed include walking distance, mobility levels, gastrointestinal function (time to first flatus and first defecation), nausea, vomiting, comfort, fatigue, time to initiation of oral intake, patient satisfaction, incidence of postoperative complications, and length of hospital stay.

Research Question:

In patients undergoing colorectal surgery (P), does a nurse-led early mobilization protocol (I), compared with standard mobilization practices (C), improve postoperative recovery outcomes (O), including walking distance, mobility levels, gastrointestinal function (time to first flatus and first defecation), nausea, vomiting, comfort, fatigue, time to initiation of oral intake, patient satisfaction, postoperative complication rates, and length of hospital stay?

DETAILED DESCRIPTION:
Colorectal surgery is a commonly performed procedure in general surgery clinics and requires intensive postoperative nursing care. Despite advances in surgical techniques, postoperative complications such as anastomotic leakage, wound infection, paralytic ileus, and pulmonary complications remain significant challenges in patients undergoing colorectal surgery.

Enhanced Recovery After Surgery (ERAS) protocols have been developed to reduce the metabolic impact of surgical stress, accelerate recovery, and decrease postoperative complications. Early mobilization is a key component of ERAS pathways and is strongly recommended within the first 24 hours following elective colorectal surgery. Early mobilization has been shown to improve gastrointestinal function, reduce postoperative fatigue, shorten hospital length of stay, and enhance overall recovery.

However, the implementation of early mobilization in routine clinical practice is often inconsistent. Institutional constraints, patient-related physical and psychological barriers, lack of knowledge, and negative beliefs regarding mobilization may delay postoperative activity, particularly in patients undergoing colorectal surgery.

Nurses play a central role in postoperative care and are well positioned to lead, coordinate, and monitor early mobilization activities. Nurse-led, structured mobilization protocols may facilitate early mobilization by providing systematic patient education, clear activity goals, and continuous monitoring during the postoperative period.

Although nurse-led mobilization protocols have been evaluated in limited randomized controlled trials across various surgical populations, evidence specifically focused on patients undergoing colorectal surgery remains scarce.

This randomized controlled trial aims to evaluate the effectiveness of a nurse-led early mobilization protocol compared with standard mobilization practices in patients undergoing elective colorectal surgery. The study focuses on postoperative recovery outcomes, including mobility, gastrointestinal function, patient comfort, fatigue, postoperative complications, patient satisfaction, and length of hospital stay. The findings of this study are expected to provide evidence to support the integration of nurse-led early mobilization protocols into routine colorectal surgical care.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Scheduled for elective colorectal surgery (e.g., procedures related to
* colorectal cancer, diverticulitis, or inflammatory bowel disease [IBD])
* Able to ambulate independently preoperatively
* Medically and cognitively able to participate in a mobilization protocol
* Able to provide written informed consent

Exclusion Criteria:

* Undergoing emergency colorectal surgery
* Patients requiring postoperative intensive care unit (ICU) admission
* Severe cognitive impairment or psychiatric disorders that may affect participation
* Musculoskeletal or neurological conditions that impair mobility
* Inability to understand study instructions due to language or communication barriers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-12-29 (Estimated); Study Completion 2026-12-29 (Estimated)

PRIMARY OUTCOMES:
Mobility level assessed | between postoperative day 0 and postoperative day 3
  Patient-reported / Observer-rated Mobility Scale The Patient Mobility Scale is used to assess pain and perceived exertion experienced during the postoperative period while performing four activities: turning from one side to the other in bed, sitting at the bedside, standing up at the bedside, and walking in the patient's room. Permission to use the scale was obtained from the responsible authors.
  The Observer Mobility Scale evaluates the degree of patient dependence/independence during mobilization activities. Blood pressure, heart rate, and respiratory rate are measured by the observer two minutes before and after mobilization.
  Furthermore, the Patient- and Observer-rated Mobility Scales will be administered on postoperative days 1, 2, and 3, and the results will be documented in the monitoring form.
Total walking distance (measured by pedometer) | between postoperative day 0 and postoperative day 3
  Mobilization will be monitored using the Mobilization Monitoring Form and step counts obtained from the pedometer will be recorded at the end of each day.
Time to first flatus (hours postoperatively) | From the end of surgery until the patient-reported first postoperative passage of flatus (within the first 72 hours postoperatively)
  The time interval (in hours) from the end of surgery to the first passage of flatus reported by the patient.
Time to first defecation (hours postoperatively) | From the end of surgery until the patient-reported first postoperative passage of defecation (within the first 72 hours postoperatively)
  The time interval (in hours) from the end of surgery to the patient's first defecation will be determined and recorded based on patient self-report.

SECONDARY OUTCOMES:
Postoperative nausea and vomiting (PONV) | during the first 3 postoperative days
  Postoperative nausea and vomiting will be assessed based on patient self-report and will be recorded by the researcher as a binary outcome (presence or absence) without using a standardized scale during the first three postoperative days.
Fatigue level | researcher during the first 3 postoperative days
  Modified Borg Scale Fatigue was assessed using the Modified Borg Scale, an 11-point scale ranging from 0 (no fatigue) to 10 (very, very hard). Patients' fatigue levels were evaluated on postoperative days 0, 1, 2, and 3.
Comfort level | Patients will be assessed on postoperative days 0, 1, 2, and 3.
  The Visual Analog Scale (VAS) is a valid, reliable, and practical measurement tool widely used to quantify subjective experiences that cannot be directly measured numerically. In this study, patient satisfaction will be assessed using the VAS (0-10). Higher VAS scores indicate greater levels of comfort.
Patient satisfaction | on postoperative day 3
  The Visual Analog Scale (VAS) is a valid, reliable, and practical measurement tool widely used to quantify subjective experiences that cannot be directly measured numerically. In this study, patient satisfaction will be assessed using the VAS (0-10). Scores ranged from 0 (low satisfaction) to 10 (high satisfaction)

CONTACTS AND LOCATIONS:
Overall Officials: Meryem N., Yavuz van Giersbergen, Study Director — Ege University
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xie, J., Luo, C., Du, Q., Zou, W., Li, X., Ma, Z., Wu, X., & Zhang, M. (2023). Factors associated with early mobilization among colorectal cancer patients after surgery: A cross-sectional study. European Journal of Oncology Nursing, 64. https://doi.org/10.1016/j.ejon.2023.102317